CLINICAL TRIAL: NCT06804616
Title: Comparison of Mucosal Vibration and Benzocaine Gel in Reducing Pain During Administration of Local Anesthesia in Children
Brief Title: Pain Reduction Using Vibration and Topical Anesthesia
Acronym: TG-EB-Eff
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UCD/ERCA/24/1108
Record Dates: First submitted 2025-01-07; First posted 2025-02-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-11

CONDITIONS: Pain Management
Keywords: Pediatric Dentistry; Pain Management; Local Anesthesia; Benzocaine Gel; Powered Toothbrush; SEM Scale; Wong-Baker Pain Scale; Pain Reduction Techniques; Randomized Control Trial
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Topical Anesthesia Group (20% Benzocaine Gel) (Active Comparator): Participants in this group will receive 20% Benzocaine Gel applied topically to the injection site for 5 minutes before administering local anesthesia. Pain levels will be assessed using both subjective (Wong-Baker FACES Pain Scale) and objective (SEM Scale) measures.
  Interventions: Drug: 20% benzocaine Gel
- Vibration Group (Powered Toothbrush) (Experimental): Participants in this group will receive vibratory stimulation using a powered toothbrush applied to the injection site for a minimum of one minute before administering local anesthesia. Pain levels will be assessed using both subjective (Wong-Baker FACES Pain Scale) and objective (SEM Scale) measures.
  Interventions: Device: Powered Toothbrush

INTERVENTIONS:
Drug: 20% benzocaine Gel — Participants in this group received 20% Benzocaine Gel applied to the injection site for 5 minutes prior to local anesthesia administration. The gel acts as a topical anesthetic to numb the area and reduce pain perception during the injection procedure.
  Other Names: Oral Anesthetic Gel, Benzocaine Oral Gel, Hurricaine Gel
  Arms: Topical Anesthesia Group (20% Benzocaine Gel)
Device: Powered Toothbrush — Participants in this group received vibration stimulation using a powered toothbrush applied to the injection site for 1 minute before the local anesthesia injection. The vibration works on the principle of gate control theory, aiming to disrupt pain signals and reduce discomfort during the injection procedure.
  Other Names: Oral-B Powered Toothbrush, Vibrating Toothbrush, Electric Toothbrush
  Arms: Vibration Group (Powered Toothbrush)

SUMMARY:
The goal of this clinical trial is to study if a powered toothbrush providing vibrations compared with 20% benzocaine topical gel is more effective in reducing pain before local anesthetic injections in children aged 6-12 years undergoing dental procedures. The main questions it aims to answer are:

Does the powered toothbrush reduce pain more effectively than the 20% benzocaine topical gel? How do children perceive and respond to each method using subjective and objective pain measurement tools?

Researchers will compare the use of a powered toothbrush to 20% benzocaine topical gel to see which method minimizes pain during infiltration anesthesia in pediatric patients.

Participants will:

Be divided into two groups:

Group A: Receive 20% benzocaine topical gel before injection. Group B: Use a powered toothbrush at the injection site before administration. Report pain levels using the Wong-Baker FACES Pain Scale and have their pain responses measured using the SEM Scale.

Study Details:

Randomized clinical trial with convenience sampling. Inclusion criteria: Children aged 6-12 years, ASA I classification, and positive Frankl behavior rating.

Exclusion criteria: Intellectual impairments, allergies to local anesthesia, or systemic health conditions.

Study duration: [November 2024 to December 2024].

Ethical Considerations:

Participation is voluntary, with informed consent required. Responses will remain confidential, and all ethical guidelines will be followed.

DETAILED DESCRIPTION:
Pain management during the administration of local anesthesia in pediatric dental patients is one of the biggest challenges in clinical practice. Pain experience can cause dental anxiety, behavioral management problems, and avoidance of necessary dental care in children. This is a randomized controlled trial of two different methods by which to diminish the perception of pain from injections of local anesthetics, namely, by the use of 20% benzocaine topical gel as a pharmacological measure and by employing a powered toothbrush as a non-pharmacological distraction technique. Investigation of these methods will provide information on their practicality and usefulness in pediatric dental environments.

Study Purpose and Rationale The overall objective of this study is to explore strategies that make dental procedures less distressing for children, ensuring better compliance, reduced anxiety, and an overall improved patient experience. Pain perception in pediatric patients is influenced by both physiological and psychological factors. Although pharmacological interventions such as benzocaine are commonly used to numb the tissue before the injection of local anesthesia, they do not deal with the anxiety or behavioral discomfort that is often associated with the injection process. In contrast, distraction techniques, especially those that incorporate vibration, can change the pain perception by breaking the transmission of pain signals and shifting the child's attention to other things.

A particularly needed contribution in the research area is therefore directly comparing the approach adopted by one or more local anaesthetics versus the benzocaine model. Although well documented in many studies about their numbing capability, the present research did not fill an important gap of comparison and competition between using the simple distraction of a vibration-powered toothbrush to reduce or prevent this severe pain upon visiting the orthodontist without much need of such a type of drug treatment or its pharmaceutical cost.

Study Design Overview

This is a randomized controlled trial. Eligible pediatric patients requiring local anesthesia for dental treatment are assigned to one of two intervention groups:

Group A (Topical Anesthetic Group): Patients in this group receive 20% benzocaine gel applied to the injection site for five minutes before the administration of local anesthesia.

Group B (Vibration Group): This group receives vibrational stimulation in the form of a powered toothbrush that is rubbed against the injection site for one minute before receiving local anesthesia.

The computerized-based randomization distributes participants evenly into the two groups to eliminate selection bias and provide an excellent comparison between interventions.

Tools of Pain Measurement

This study makes use of two valid tools that assess the patient's pain perception:

SEM Scale: This is an observational tool that is used to measure pain-related behaviors during the injection process. It measures the child's vocal responses (sound), eye movements, and motor reactions, providing a composite score that reflects their pain-related behavior.

Wong-Baker FACES Pain Scale: This self-report measure is taken as the child assesses the severity of pain that occurred after receiving the injection. A series of images of facial expressions representing "no pain" through "worst pain" are used, which children then assign a number score.

The above two tools integrate to capture both objective and subjective measurements of pain; therefore, a comprehensive analysis is achieved by evaluating the effectiveness of each intervention.

Intervention Procedures Each intervention is administered immediately before the injection of local anesthesia (2% lidocaine with epinephrine). The procedures are standardized and carried out by a single trained dentist to ensure consistency across participants. This approach minimizes variability and ensures that the outcomes accurately reflect the differences between the interventions.

Study Population and Inclusion Criteria Participants are pediatric patients aged 6 to 12 years requiring local anesthesia for dental procedures.

Patients categorized as ASA Class I, i.e., patients who are healthy. No allergic history of the patient to topical anesthetics and any other materials used in this study.

Patient behavior was graded as positive or definitely positive based on the Frankl Behavior Rating Scale (3 and 4 scores).

Exclusion criteria include systemic complications, severe dental anxiety or phobia, or active oral/systemic infections. These criteria ensure the safety of participants and the reliability of the study results.

Ethical Considerations The study follows the principles of the Declaration of Helsinki and is approved by the appropriate institutional ethics review board. Informed consent is sought from the parents or guardians of all participants.

Significance of the Study This trial is of great significance to pediatric dental practice. If this powered toothbrush is proven as effective as benzocaine gel in pain perception, it will be a cheap, non-invasive alternative to pharmacological agents, especially where such agents may not be easily accessible. Besides, the method of distraction addresses the physical and psychological aspects of pain, thus decreasing dental anxiety and improving compliance with the patient.

By basing evidence on recommendations from this study, improving quality care is hoped to provide a more quality life for these children and promote innovation in applying the patient-friendlier method of techniques at clinical levels.

Data Analysis: Statistical analyses will be performed to compare pain scores between the two groups. Descriptive statistics will summarize demographic and baseline characteristics, while inferential tests such as t-tests or ANOVA will assess differences in SEM and Wong-Baker scale scores.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years.
* Children classified as ASA I (American Society of Anesthesiologists).
* Children with FRANKL Behavior Rating Scale of "positive" or "definitely positive."

Exclusion Criteria:

* Intellectually impaired/Autistic
* Patient allergic to L.A
* Patient with systemic health condition

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Measure Title: Pain Levels as Assessed by SEM (Sound, Eye, Motor) Scale | "During the intervention, within 5 minutes"
  Evaluation of objective pain responses during local anesthesia administration using the SEM scale. Scores range from 0 (no pain) to 9 (severe pain).
Pain Levels as Assessed by Wong-Baker FACES Pain Scale | "Immediately after the intervention, within 1-5 minutes"
  Self-reported subjective pain levels assessed by the Wong-Baker FACES scale, ranging from 0 (no hurt) to 10 (hurts worst).

CONTACTS AND LOCATIONS:
Overall Officials: Irsam Haider, BDS, MCPS, Principal Investigator — University of Lahore
Locations (1):
- University Of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study will not be shared with other researchers to protect the confidentiality and privacy of the participants. Since the study involves pediatric patients, maintaining strict adherence to ethical guidelines and ensuring data security is paramount. Furthermore, the scope of this study is limited to internal analysis, and no provisions for external data sharing were included in the consent obtained from participants or their guardians

REFERENCES:
- [Background] AlHareky M, AlHumaid J, Bedi S, El Tantawi M, AlGahtani M, AlYousef Y. Effect of a Vibration System on Pain Reduction during Injection of Dental Anesthesia in Children: A Randomized Clinical Trial. Int J Dent. 2021 Jan 30;2021:8896408. doi: 10.1155/2021/8896408. eCollection 2021. PMID 33564311
- [Background] Shilpapriya M, Jayanthi M, Reddy VN, Sakthivel R, Selvaraju G, Vijayakumar P. Effectiveness of new vibration delivery system on pain associated with injection of local anesthesia in children. J Indian Soc Pedod Prev Dent. 2015 Jul-Sep;33(3):173-6. doi: 10.4103/0970-4388.160343. PMID 26156269
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Shaefer JR, Lee SJ, Anderson NK. A Vibration Device to Control Injection Discomfort. Compend Contin Educ Dent. 2017 Jun;38(6):e5-e8. PMID 28586233
- See also: Vibrating toothbrush, ice, or topical anesthetic agent to reduce pain of local anesthetic injection in 5- to 12-year-old children undergoing dental procedures - a randomized controlled trial — https://journals.ekb.eg/article_329890.html
- See also: Comparison of Three Different Techniques to Allay Anxiety before Local Anesthesia Injection in Pediatric Population — http://edelweisspublications.com/edelweiss/article/comparison-three-different-techniques-allay-anxiety-local-anesthesia-2572-6978-drm-19-127.pdf